CLINICAL TRIAL: NCT05712759
Title: Surveillance of Nosocomial Influenza at Edouard Herriot University Hospital, Lyon, France
Brief Title: Nosocomial Influenza Surveillance of 2022 - 2027 Seasonal Period
Acronym: NOSOGRIPPE
Status: Withdrawn | Type: Observational
Why Stopped: change of study design
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_1064
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Infection Viral
Keywords: influenza; hospital; nosocomial
MeSH Terms: conditions — Virus Diseases; Influenza, Human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Influenza-like illness group — Each patient who present ILI (influenza-like illness) at admission or during hospitalization and who have had a nasopharyngeal swab taken as part of their care for the purpose of diagnosing influenza by Polymerase Chain reaction (PCR) testing.
  ILI is defined by fever > 37,8°C or/and cough or sore throat.

SUMMARY:
Hospital-Acquired Influenza (HAI) is closely linked to the intensity of influenza in the community. HAI is associated with significant morbidity, mortality and extra costs due to prolonged hospital stay. The incidence of laboratory confirmed HAI has been reported rarely. The proportion of HAI among influenza cases was 11.38% (95% Confidence Interval: 5.19%-19.55%) in a meta-analysis of 14 studies. In France, a prospective surveillance study of adults with Influenza-Like Illness (ILI) over 11 years, reported that 35.6% of the influenza cases diagnosed at hospital were hospital-acquired.

HAI is transmitted via respiratory droplets and by hand contacts. The spread is facilitated by Health Care Professionals (HCPs), patients and visitors.

Prevention and control of HAI is of upmost importance to preserve patient safety and limit the related economic costs. While vaccination of HCPs has been shown to contribute to the reduction of HAI, less is known on the impact of patient vaccination on the risk of HAI during hospitalization.

The aim of this study is to describe the hospital-acquired influenza in a french university hospital.

ELIGIBILITY:
Inclusion Criteria:

* Any volunteer adult patient (≥ 18 years of age) hospitalized for at least 24 hours on a study unit, who had a nasopharyngeal swab taken as part of care for the purpose of diagnosing influenza by PCR testing and who had an influenza-like illness meeting the following definition:
* Fever greater than 37.8°C in the absence of antipyretics; And/or
* Cough or pharyngeal pain.

Exclusion Criteria:

* Any person who does not meet the above definition or who has expressed opposition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any volunteer adult patient (≥ 18 years of age) hospitalized at Edouard Herriot Hospital for at least 24 hours on a study unit, who had a nasopharyngeal swab taken as part of care for the purpose of diagnosing influenza by PCR testing and who had an influenza-like illness meeting the following definition
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-03-09 (Actual); Primary Completion 2025-03-09 (Actual); Study Completion 2025-03-09 (Actual)

PRIMARY OUTCOMES:
To describe and document cases of nosocomial influenza occurring at Edouard Herriot Hospital. | At inclusion
  The primary endpoint will be assessed by the proportion of patients with nosocomial influenza among all patients with influenza-like illness during an influenza season.